CLINICAL TRIAL: NCT01564277
Title: Efficacy and Safety of Two Comparable Single Low Doses of Rasburicase Followed by Allopurinol in Adult Patients With Malignancy
Brief Title: Rasburicase and Allopurinol in Treating Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 197711; NCI-2011-03231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 197711 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-27 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; de Novo Myelodysplastic Syndromes; Noncontiguous Stage II Adult Burkitt Lymphoma; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Stage I Adult Burkitt Lymphoma; Stage III Adult Burkitt Lymphoma; Stage IV Adult Burkitt Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma | interventions — rasburicase; Peplomycin; Urate Oxidase; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (1.5mg rasburicase) (Experimental): Patients receive 1.5mg of rasburicase IV over 30 minutes on day 1 and allopurinol PO QD on days 1-6.
  Interventions: Drug: rasburicase; Drug: allopurinol
- Arm II (3 mg rasburicase) (Experimental): Patients receive 3 mg of rasburicase IV over 30 minutes on day 1 and allopurinol PO QD on days 1-6.
  Interventions: Drug: rasburicase; Drug: allopurinol

INTERVENTIONS:
Drug: rasburicase — Given IV
  Other Names: Elitek; NK-631; recombinant urate oxidase
Drug: allopurinol — Given PO
  Other Names: 4'-HPP; ALLO; Zyloprim

SUMMARY:
This randomized phase II trial studies how well giving rasburicase together with allopurinol works in treating patients with hematologic malignancies. Rasburicase may reduce the level of uric acid in the blood. Allopurinol may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known which dose of rasburicase is more effective in treating hematologic malignancies when given together with or without allopurinol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively evaluate the efficacy, as defined by uric acid response rate, of 2 different single low doses of rasburicase followed by allopurinol in 2 treatment arms.

SECONDARY OBJECTIVES:

I. To estimate the proportion of patients requiring additional doses of rasburicase to maintain a uric acid level =< 7.5mg/dL on day 2 through day 6.

II. To identify differential characteristics of the patients who do not respond to treatment.

III. To measure the area under the plasma uric acid concentration-time curve (AUC) from baseline (day 1) to day 7, time to plasma uric acid level less than or equal to 7.5mg/dL.

IV. To evaluate the rate of patients requiring hemodialysis (HD) V. To evaluate the safety of low single-doses of rasburicase. VI. To evaluate the rate of patients expressing a doubling of serum creatinine.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive 1.5mg of rasburicase intravenously (IV) over 30 minutes on day 1* and allopurinol orally (PO) once daily (QD) on days 1-6.

ARM II: Patients receive 3 mg of rasburicase IV over 30 minutes on day 1* and allopurinol PO QD on days 1-6.

NOTE: *Patients with serum uric acid >= 7.5mg/dl also receive rasburicase IV on days 2-3.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status of 0-3
* Active leukemia and Burkitt leukemia/lymphoma treated in-house that puts them at risk for tumor lysis syndrome (TLS)
* Serum uric acid level >= 7.5mg/dL and high risk for TLS as defined by:

  * A diagnosis of acute myeloid leukemia (AML), or
  * A diagnosis of blast-phase chronic myeloid leukemia (CML), or
  * A diagnosis of high-grade myelodysplastic syndrome (MDS) with >= 10% blast bone marrow blast involvement, or
  * Acute lymphoblastic leukemia (ALL), or
  * Burkitt leukemia/lymphoma
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* History of asthma
* History of severe or life threatening atopic allergy
* Hypersensitivity to uricases
* Known prior sensitivity to allopurinol
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Recent prior history of uricolytic therapy defined as therapy within the last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09-29 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2016-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Wang, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.5) | 68.4 (16.4) | 69.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Probability of Obtaining a Uric Acid Level =< 7.5mg/dL
Description: The proportion of patients able to achieve and/or maintain a uric acid level =< 7.5mg/dL for each treatment arm.
Time Frame: Within 24 hours of rasburicase treatment
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
proportion of participants | 0.83 [0.52 to 0.98] | 0.67 [0.35 to 0.90]

2. Secondary Outcome: Number of Patients Requiring Additional Doses of Rasburicase to Maintain a Uric Acid Level =< 7.5mg/dL
Description: Count of partcicpants requiring additional doses of rasburicase to maintain a uric acid level =< 7.5mg/dL by treatment arm.
Time Frame: Up to day 7
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
Participants | 1 | 3

3. Secondary Outcome: Baseline White Blood Cell Count by Response
Description: The mean baseline white blood cell count of patients with a complete response (CR) (patients who achieved uric acid level =< 7.5mg/dL) and no CR (patients with uric acid level > 7.5mg/dL).
Time Frame: Up to day 7
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
cells x 10^9/L
  Complete Response: number analyzed (Participants) | 10 | 8
  Complete Response | 62.1 (32.3) | 29.0 (34.0)
  No Complete Response: number analyzed (Participants) | 2 | 4
  No Complete Response | 13.9 (17.1) | 33.3 (19.0)

4. Secondary Outcome: Area Under the Plasma Uric Acid Concentration-time Curve (AUC) From Baseline (Day 1) to Day 7
Description: The mean area under the plasma uric acid concentration-time curve (AUC) from baseline (Day 1) to Day 7
Time Frame: Up to day 7
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: days*mg/dL
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
days*mg/dL | 12.5 (9.0) | 3.5 (4.7)

5. Secondary Outcome: Safety of Low Single-doses of Rasburicase.
Description: The number of patients with any adverse events .
Time Frame: up to day 7
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

6. Secondary Outcome: Number of Patients Experiencing a Doubling of Serum Creatinine
Description: Count of participants experiencing a doubling of serum creatinine
Time Frame: up to day 6
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (1.5mg Rasburicase) | Arm II (3 mg Rasburicase)
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (1.5mg Rasburicase) (N=12) | Arm II (3 mg Rasburicase) (N=12)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (1.5mg Rasburicase) (N=12) | Arm II (3 mg Rasburicase) (N=12)
Anaemia (Blood and lymphatic system disorders) | 6 (38) | 4 (10)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (8) | 2 (8)
Leukopenia (Blood and lymphatic system disorders) | 7 (44) | 4 (14)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 6 (44) | 3 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (54) | 5 (14)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (2)
Cushingoid (Endocrine disorders) | 1 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (12) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 8 (16) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 2 (4)
Proctalgia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (4)
Asthenia (General disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (6) | 3 (6)
Malaise (General disorders) | 2 (4) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2)
Oedema (General disorders) | 4 (10) | 0 (0)
Oedema peripheral (General disorders) | 3 (6) | 5 (14)
Pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 2 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (8) | 2 (6)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Candidiasis (Infections and infestations) | 1 (2) | 1 (2)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (2)
Herpes virus infection (Infections and infestations) | 1 (2) | 0 (0)
Mastitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (8) | 2 (4)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Chemical eye injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound secretion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (10) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 1 (8) | 5 (10)
Blood alkaline phosphatase increased (Investigations) | 1 (4) | 3 (10)
Blood bilirubin increased (Investigations) | 2 (4) | 4 (12)
Blood creatinine (Investigations) | 0 (0) | 2 (4)
Blood creatinine increased (Investigations) | 3 (12) | 2 (8)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (2)
Breath sounds (Investigations) | 1 (2) | 0 (0)
Haemoglobin (Investigations) | 2 (6) | 2 (8)
Lymphocyte count decreased (Investigations) | 5 (30) | 2 (10)
Neutrophil count decreased (Investigations) | 1 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (8) | 2 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (4) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (6) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (28) | 6 (20)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (44) | 8 (32)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (12) | 6 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (6) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (12) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 2 (4) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6)
Catheter removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Embolism (Vascular disorders) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 2 (4)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 2 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes